CLINICAL TRIAL: NCT06635148
Title: Long-term Extension Study for Participants With Geographic Atrophy (GA) Secondary to Age-related Macular Degeneration (AMD) in JNJ-81201887 Parent Clinical Studies
Brief Title: A Long-term Extension Study of JNJ-81201887 (AAVCAGsCD59) Parent Studies in Participants With Geographic Atrophy (GA) Secondary to Age-related Macular Degeneration (AMD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81201887MDG3002; 81201887MDG3002 (Other: Janssen Research & Development, LLC); 2022-500747-21-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-09-23; First posted 2024-10-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Geographic Atrophy; Macular Degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Long-term safety study of a single intravitreal dose of JNJ-81201887 administered during parent studies (81201887MDG2001: Randomized trial; 81201887MDG1003: Non-randomized trial)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: JNJ-81201887 Low Dose (Experimental): Study participants who were enrolled and received treatment with low dose JNJ-81201887 in parent clinical studies (81201887MDG2001 [NCT05811351]; 81201887MDG1003) will enter this long-term extension (LTE) study. No study intervention will be administered as part of this study.
  Interventions: Drug: JNJ-81201887
- Arm B: JNJ-81201887 High dose (Experimental): Study participants who were enrolled and received treatment with high dose JNJ-81201887 in parent clinical studies (81201887MDG2001 [NCT05811351]; 81201887MDG1003) will enter this LTE study. No study intervention will be administered as part of this study.
  Interventions: Drug: JNJ-81201887
- Arm C: Sham Procedure (Sham Comparator): Participants randomized to the sham arm in parent study 81201887MDG2001 (NCT05811351) may have the option to receive JNJ-81201887 open-label treatment under a separate protocol after unmasking of that study; and will enter this LTE study. No intervention will be administered as part of this study.
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Drug: JNJ-81201887 — No study intervention will be administered as part of this LTE study.
  Arms: Arm A: JNJ-81201887 Low Dose; Arm B: JNJ-81201887 High dose
Other: Sham Procedure — No study intervention will be administered as part of this LTE study.
  Arms: Arm C: Sham Procedure

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability after an intravitreal injection (a shot of medicine into the eye) of JNJ-81201887 administered in parent clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were enrolled and received treatment with JNJ-81201887 or sham in a parent clinical study (81201887MDG2001, 81201887MDG1003)
* Females (women of childbearing potential), male participants, and partners of male participants will not be required to use contraception in this LTE study
* Must sign an informed consent form (ICF) indicating that participant understands the purpose of, and procedures required for, the study and is willing to participate in the study. The ICF may be signed by an impartial witness and/or legally designated representative depending on national/local regulations

Exclusion Criteria:

* There are no exclusion criteria for this LTE study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2029-08-24 (Estimated); Study Completion 2030-06-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Ocular and Systemic Treatment-emergent Adverse Events (TEAEs) | Upto 5 Years
  Number of participants with ocular and systemic TEAEs will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as any adverse event occurring at or after the administration of study intervention.
Number of Participants with Abnormal Findings in Clinical Laboratory Assessments | Upto 5 Years
  Number of participants with abnormal findings in clinical laboratory Assessments (including hematology and clinical chemistry) will be reported.
Number of Participants with Abnormal Findings in Retinal imaging and Eye Examinations | Upto 5 Years
  Number of participants with abnormal findings in retinal imaging (Fundus Autofluorescence, Spectral Domain Optical Coherence Tomography, Color Fundus Photography) and eye examinations will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (104):
- United States (46):
  - Retina Associates Southwest PC, Tucson, Arizona
  - Retina Consultants of Orange County, Fullerton, California
  - Shiley Eye Institute Jacobs Retina Center, La Jolla, California
  - California Retina Consultants, Oxnard, California
  - California Eye Medical Specialists, Pasadena, California
  - Retina Consultants San Diego, Poway, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Group of Florida, Fort Lauderdale, Florida
  - VitreoRetinal Associates, PA, Gainesville, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Georgia Retina, Marietta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - University Retina, Lemont, Illinois
  - Midwest Eye Institute, Carmel, Indiana
  - Maine Eye Center, Portland, Maine
  - Retina Specialists, Baltimore, Maryland
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Retina Consultants of Minnesota, Saint Louis Park, Minnesota
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Retina-Vitreous Surgeons of Central New York, Liverpool, New York
  - Asheville Eye Associates - Western Carolina Retinal Associates, Asheville, North Carolina
  - Duke Eye Center, Durham, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - NC Retina Associates, Wake Forest, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Verum Research LLC, Eugene, Oregon
  - Cascade Medical Research Institute, LLC, Springfield, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Charleston Neuroscience Institute, LLC, Beaufort, South Carolina
  - Austin Clinical Research, Austin, Texas
  - Retina and Vitreous of Texas, PLLC, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Retina Associates Of South Texas P A, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group, Willow Park, Texas
  - University of Utah, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Research institute, Norfolk, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
- Australia (4):
  - Centre for Eye Research Australia, East Melbourne
  - Strathfield Retina Clinic, Strathfield
  - Sydney Retina Clinic and Day Surgery, Sydney
  - Sydney West Retina, Westmead
- Belgium (3):
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Alberta Retina Consultants, Edmonton, Alberta, Canada
- China (3):
  - Beijing Tongren Hospital CMU, Beijing
  - West China Hospital Si Chuan University, Chengdu
  - Shanghai General Hospital, Shanghai
- Czechia (2):
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - AXON Clinical s.r.o., Prague
- University Hospital Of Copenhagen, Glostrup Hospital, Glostrup Municipality, Denmark
- Germany (7):
  - Universitaets-Augenklinik Bonn, Bonn
  - Klinikum Gottingen der Georg August Universitat, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum Ludwigshafen, Ludwigshafen am Rhein
  - Augenzentrum am St Franziskus Hospital Munster, Münster
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (3):
  - Eszak Pesti Centrumkorhaz Honvedkorhaz, Budapest
  - Ganglion Orvosi Központ, Pécs
  - Zala Varmegyei Szent Rafael Korhaz, Zalaegerszeg
- Italy (6):
  - Azienda Ospedaliero Universitaria di Ferrara, Ferrara
  - ASST Fatebenefratelli Sacco, Milan
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Luigi Vanvitelli, Napoli
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
- Netherlands (2):
  - Radboudumc, Nijmegen
  - Het Oogziekenhuis Rotterdam, Rotterdam
- Poland (2):
  - Oftalmika, Bydgoszcz
  - Warszawski Szpital Okulistyczny, Warsaw
- Portugal (3):
  - Uls Coimbra - Hosp. Univ. Coimbra, Coimbra
  - Espaco Medico de Coimbra, Coimbra
  - Uls Sao Joao, Porto
- Spain (13):
  - Centro de Oftalmologia Barraquer, Barcelona
  - Centro Medico Teknon S.L., Barcelona
  - Inst. Cat. de Retina, Barcelona
  - Clinica Oftalvist Valencia, Burjassot
  - Hosp. La Arruzafa, Córdoba
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Baviera Madrid Castellana, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Clinica Univ. de Navarra, Pamplona
  - Idc Salud Hosp. Gral. de Catalunya, Sant Cugat del Vallès
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
- S:t Eriks Ogonsjukhus, Stockholm, Sweden
- Inselspital Universitatsspital Bern, Bern, Switzerland
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Ankara
  - Baskent University Ankara Hospital, Ankara
- United Kingdom (4):
  - Bristol Eye Hospital, Bristol
  - Oxford Eye Hospital, Headington
  - The Retina Clinic London, London
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency